CLINICAL TRIAL: NCT04365764
Title: Effect of Treatments in Patients Hospitalized for Severe COVID-19 Pneumonia: a Multicenter Cohort Study
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Centre Hospitalier Intercommunal Robert Ballanger (Other); Centre Hospitalier Intercommunal Montfermeil-Le Raincy (Unknown); CMC Ambroise Paré (Other)
Responsible Party: Principal Investigator, Lee S Nguyen, Study coordinator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-20-06
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Covid-19; ARDS; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed to the treatment: Exposure variable will be studied treatment
- Not exposer to the treatment (control group)

SUMMARY:
Several treatments have been used in during the Covid-19 pandemic of 2020. Using patients' registries from several hospitals in Paris, the investigators retrospectively analyzed associations between specific treatments, including but not limited to vaccines targeted against SARS-CoV-2, hydroxychloroquine, azithromycin, remdesivir, baricitinib, tocilizumab, sarilumab, lopinavir/ritonavir and oseltamivir; and clinical outcomes including, death and mechanical ventilation.

DETAILED DESCRIPTION:
Several treatments have been used in during the Covid-19 pandemic of 2020. Using patients' registries from several hospitals in Paris, the investigators retrospectively analyzed associations between specific treatments, including but not limited to vaccines targeted against SARS-CoV-2, hydroxychloroquine, azithromycin, remdesivir, baricitinib, tocilizumab, sarilumab, lopinavir/ritonavir and oseltamivir; and clinical outcomes including, death and mechanical ventilation.

Other outcomes of interest include: acute kidney injury, encephalopathy, need for intensive care unit transfers.

ELIGIBILITY:
Inclusion Criteria:

* admitted for severe Covid-19 pneumonia (i.e. requiring O2-support more than 6L/min with SpO2<96%)

Exclusion Criteria:

* patients who were previously in ICU
* patients already hospitalized prior to study start date
* patients in palliative care
* lack of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is cohort-base in routine care, in medical departments.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-03-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Composite of death and mechanical ventilation | 14-days follow-up
  Composite of death and mechanical ventilation (i.e. intubation)

SECONDARY OUTCOMES:
Death | 14-days follow-up
  Death
Mechanical ventilation | 14-days follow-up
  Enabled by intubation
Composite of death and mechanical ventilation | 28-days follow-up
  Composite of death and mechanical ventilation
World Health Organization score | 14-days follow-up
  World Health Organization score
World Health Organization score | 28-days follow-up
  World Health Organization score

CONTACTS AND LOCATIONS:
Overall Officials: Joe-Elie Salem, MD, PhD, Study Chair — APHP
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier Intercommunal Le Raincy-Montfermeil, Montfermeil

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be available on request.